CLINICAL TRIAL: NCT00232479
Title: Phase II Study of Dose Dense Carboplatin and Taxotere With Herceptin As Primary Systemic Therapy in Breast Cancer
Brief Title: Dose Dense Carboplatin, Taxotere and Herceptin As Primary Systemic Therapy in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Judith Hurley, MD, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC 2004-064
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm 1 (Experimental): single arm study evaluating the efficacy of neoadjuvant taxotere, herceptin and carboplatin given in a dose dense fashion
  Interventions: Drug: trastuzumab, docetaxel and carboplatin in dose dense regimen

INTERVENTIONS:
Drug: trastuzumab, docetaxel and carboplatin in dose dense regimen — trastuzumab 4 mg/kg day 1 and then 2 mg/kg/week x 11, carboplatin 6 mg AUC Day 1, 15, 29, 43, docetaxel 75 mg/meter squared Days 1, 15, 29, 43, neulasta 6 mg Day 2, 16, 30, 44
  Other Names: herceptin, taxotere and carboplatin

SUMMARY:
Dose dense therapy has been shown to increase survival in the adjuvant setting of breast cancer. It is unknown if dose dense therapy will improve survival in tumors that express her-2. This study evaluates a neoadjuvant regimen containing carboplatin, taxotere and herceptin when used in a dose dense manner in patients with large breast cancers. The endpoint of pathologic complete response is used as a surrogate marker for survival.

DETAILED DESCRIPTION:
Dose dense therapy has been shown to increase survival in the adjuvant setting of breast cancer. It is unknown if dose dense therapy will improve survival in tumors that express her-2. This study evaluates a neoadjuvant regimen containing carboplatin, taxotere and herceptin when used in a dose dense manner in patients with large breast cancers. The endpoint of pathologic complete response is used as a surrogate marker for survival.Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations

ELIGIBILITY:
Inclusion Criteria:

* HER-2 overexpressing breast cancer
* Clinical stage 2-3B
* Normal ejection fraction

Exclusion Criteria:

* Metastatic disease
* Low ejection fraction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hurley, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: study group receives taxotere, herceptin and carboplatin in dose dense fashion
Period: Overall Study
Arm/Group | Group 1
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: treat with taxotere, herceptin, carboplatin in dose dense fashion
Arm/Group | Group 1
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathologic Complete Response (pCR)
Description: pCR is defined as the absence of invasive tumor from the surgical specimen of breast and axilla which is obtained after the chemotherapy regimen has been delivered.
Time Frame: determined at the time of surgery which is approximately 16 weeks from the beginning of treatment
Population: 48 patients signed consent but only 44 were evaluable. To be evaluable the patient must have received at least one dose of chemo and then had surgery. Two patients withdrew consent before treatment and two patients did not have surgery. So 44 are evaluable for the primary endpoint
Measure: Number; unit: participants
Groups:
- Group 1: patients received dose dense herceptin, carboplatin and taxotere
Arm/Group | Group 1
Number analyzed (Participants) | 44
participants | 19

2. Secondary Outcome: Safety and Tolerability
Description: the number of patients with grade 4 (severe) toxicities and or hospitalizations were measured to assess safety and tolerability
Time Frame: from the first dose of chemotherapy until surgery which was approximately 16 weeks.
Population: 48 patients signed an initial informed consent. 2 withdrew consent before treatment. 2 withdrew after starting treatment. Only 44 are evaluable for primary endpoint because 2 did not go for surgery.
Measure: Number; unit: participants
Groups:
- Group 1: patients received herceptin, carboplatin and taxotere in a dose dense fashion.
Arm/Group | Group 1
Number analyzed (Participants) | 44
participants | 1

ADVERSE EVENTS:
Time Frame: adverse events were collected for the 16 week pre-operative period while the study was open to accrual over a three year period.
Description: toxicity coded and graded using the CTC 2.0
Groups:
- Group 1: patients received herceptin, carboplatin, taxotere in dose dense fashion
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=46)
hospitalization (Gastrointestinal disorders) | 1 (1) — one patient hospitalized for nausea, vomiting, diarrhea and dehydration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less